CLINICAL TRIAL: NCT06704438
Title: Diagnostic and Prognostic Value of D-Lactate and Scube-1 Levels in Critically Ill Patients
Status: Completed | Type: Observational
Sponsor: Kanuni Sultan Suleyman Training and Research Hospital (Other)
Responsible Party: Principal Investigator, Ramiz Yazıcı, ASISTANT PROFESSOR, Kanuni Sultan Suleyman Training and Research Hospital
Other Study IDs: 2019/17348
Record Dates: First submitted 2024-11-21; First posted 2024-11-26 (Actual); Last update posted 2024-11-26 (Actual); Status verified 2024-11

CONDITIONS: Critical Illness; D-Lactate; SCUBE-1
Keywords: D-Lactate; SCUBE-1; Critical Illness
MeSH Terms: conditions — Critical Illness

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Control Group: The control group consisted of healthy individuals without any disease who voluntarily participated in the study.
  Interventions: Diagnostic Test: D-Lactate
- Patients Group: Patients over the age of 18 who were diagnosed as critically ill by the emergency department physician and who gave informed consent were included in the study.
  Interventions: Diagnostic Test: D-Lactate

INTERVENTIONS:
Diagnostic Test: D-Lactate — D-Lactate and SCUBE-1 can be used as early diagnosis and mortality indicators in critically ill patients.

SUMMARY:
The investigators aimed to investigate the diagnostic and prognostic levels of D-Lactate and SCUBE-1 in critically ill patients being admitted to the emergency department.

DETAILED DESCRIPTION:
Patients who were diagnosed according to the criteria as being critically ill by the ED responsible physician (patients whose basic vital functions are unstable, who receive supportive treatment or whose general condition is expected to deteriorate) were included. Patients over 18 years of age who agreed to participate in the study were included after consent was obtained from the patient or their relatives. Patients who did not meet the definition of critical patients, whose follow-up was incomplete, who did not want to participate in the study, pregnant women, and patients under 18 years of age were all excluded. A healthy control group was formed from the relatives of the patients who came to the ED outpatient clinics, as well as hospital staff who wanted to participate in the study.

Age, gender, known diseases, medications, vital parameters, and the laboratory results from critically ill patients and healthy volunteers admitted to the ED were recorded, and blood samples taken for D-Lactate and SCUBE-1 at the time of admission to the emergency room were placed in Ethylenediaminetetraacetic acid (EDTA) tubes. Clinical scores, such as the Glasgow Coma Scale (GCS), Acute Physiology and Chronic Health Evaluation (APACHE) II, Revised Trauma Score (RTS), and shock index were calculated. Critical patients were divided into the following seven groups according to their emergency department diagnosis: central nervous system, cardiovascular system, respiratory system, gastrointestinal system/metabolic, sepsis, trauma, and other. The clinical outcomes of these patients (ED length of stay, ICU or ward admission, ED and ICU mortality) were also noted. The relationship between the patient's clinical scoring (GCS, APACHE II, RTS and shock index ), laboratory results, and mortality status with D-Lactate and SCUBE-1 levels was compared. At the same time, the diagnostic value of d-lactate and SCUBE-1 for distinguishing critically ill patients was investigated.

ELIGIBILITY:
Inclusion Criteria:

Age 18 years or older Evaluated as critically ill by emergency department physician

Exclusion Criteria:

Patients not meeting critical illness criteria Patients with incomplete follow-up records Patients who declined to participate in the study Pregnant women Individuals under 18 years of age

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients who were diagnosed according to the criteria as being critically ill by the ED responsible physician (patients whose basic vital functions are unstable, who receive supportive treatment or whose general condition is expected to deteriorate) were included. Patients over 18 years of age who agreed to participate in the study were included after consent was obtained from the patient or their relatives. Patients who did not meet the definition of critical patients, whose follow-up was incomplete, who did not want to participate in the study, pregnant women, and patients under 18 years of age were all excluded. A healthy control group was formed from the relatives of the patients who came to the ED outpatient clinics, as well as hospital staff who wanted to participate in the study. Critical patients were divided into the following seven groups according to their emergency department diagnosis: central nervous system, cardiovascular system, respiratory system, gastrointestinal syst
Sampling Method: Non-Probability Sample
Enrollment: 90 (Actual)
Dates: Start 2019-07-25 (Actual); Primary Completion 2020-01-01 (Actual); Study Completion 2020-01-15 (Actual)

PRIMARY OUTCOMES:
Comparison of D-Lactate and SCUBE-1 levels in patients who were diagnosed according to the criteria as being critically ill by the ED responsible physician and a control group | The study was conducted with blood samples taken at the time of admission. The outcome measure will be assessed up to 24 weeks.
  The investigators compared the plasma blood levels of biomarkers in both groups

CONTACTS AND LOCATIONS:
Locations (1):
- Kanuni SUltan Suleyman Training and Research Hospital, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
It can be shared upon reaching the corresponding author.

REFERENCES:
- [Background] Mitarai T, Gordon AJ, Nudelman MJR, Urdaneta AE, Nesbitt JL, Niknam K, Graber-Naidich A, Wilson JG, Kohn MA. Association of an Emergency Critical Care Program With Survival and Early Downgrade Among Critically Ill Medical Patients in the Emergency Department. Crit Care Med. 2023 Jun 1;51(6):731-741. doi: 10.1097/CCM.0000000000005835. Epub 2023 Apr 3. PMID 37010317
- [Background] Tahirli T, Altuncı YA, Yalçınlı S. The Evaluation of In-Hospital Transportation of Emergency Room Critically Ill Patients. Genel Tıp Derg
- [Background] Robertson LC, Al-Haddad M. Recognizing the critically ill patient. Anaesthesia & Intensive Care Medicine